CLINICAL TRIAL: NCT00297024
Title: MRI Changes With Administered Oxygen and Carbon Dioxide in Patients With Brain Tumors Receiving Radiotherapy: A Pilot Study
Brief Title: Radiotherapy - Cerebrovascular Reactivity (RT-CVR Study)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHN REB 04-0750-C
Record Dates: First submitted 2006-02-23; First posted 2006-02-27 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2014-01

CONDITIONS: Brain Neoplasms
MeSH Terms: conditions — Brain Neoplasms

ARMS (1):
- MRI for brain mets (Experimental)
  Interventions: Procedure: MRI

INTERVENTIONS:
Procedure: MRI — Patients will be scanned while breathing in varying amounts of oxygen and carbon dioxide in varying amounts through a breathing device.

SUMMARY:
Brain tumours often have low oxygen levels, and that makes them more resistant to radiation therapy. If patients breathe the right mixture of oxygen during treatment, radiation may work better. In this study, patients with brain tumour will undergo a special MRI test while they breathe different mixtures of oxygen and carbon dioxide to find out whether oxygen levels improve in the tumor. Patients will also be asked to repeat this MRI test during the second week of radiation therapy, as well as 3 months, 6 months and 1 year after RT. The MRI test after RT will help us understand how the blood vessels in the normal brain are affected by radiation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary gliomas visible on MRI who are planning to receive radiotherapy or
* Patients with brain metastases>1cm who are planning to receive radiotherapy
* Karnofsky Performance Status >60
* Age 18 years
* Patients must be willing to visit Toronto Western Hospital for at least one MRI scan prior radiotherapy

Exclusion Criteria:

* Seizures not controlled with medications, or non compliance with prescribed anti-seizure medication
* Prior radiation therapy to the brain
* Pregnancy
* Unwilling or unable to co-operate with breathing maneuvers
* Respiratory or cardiac limitations to breathing at 20 L/min
* Medical contra-indications to limited hypercapnia or hypocapnia (known increased intracerebral pressure, metabolic acidosis or alkalosis)
* Contraindication to MRI (patients weighing>136 kgs-weight limit for the scanner tables; allergy to MR contrast agent; patients with pacemakers, cerebral aneurysm clips, shrapnel injury or implantable electronic devices not compatible with MRI)
* Other medical conditions deemed by the PI or associates to make the patients ineligible for protocol procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2005-02; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
- To measure the inter-patient variability of change in tumour oxygenation with carbogen adminstration using MRI | 2 years

SECONDARY OUTCOMES:
- To determine whether modulation of oxygen and carbon dioxide administration can improve tumour oxygenation relative to standard carbogen breathing on MRI | 2 years
- To determine whether changes in tumour oxygenation with carbogen administration are different during the second week of radiotherapy compared to baseline measurements | 2 years
- To determine whether the normal brain cerebrovascular reactivity (CVR) measured with MRI changes through a course of radiotherapy and follow-up | 2 years
- To determine whether CVR differs between radiation exposed and non-exposed normal brain tissue in a given patient after radiotherapy | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Ménard, MD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- University Health Network, Toronto, Ontario, Canada